CLINICAL TRIAL: NCT01596231
Title: Isoflavone (Kudzu) Extract Effects on Alcohol Drinking: Single Dose Pretreatment Study
Brief Title: Kudzu Treatment for Alcohol Abuse
Acronym: KUDZU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Scott Lukas, Director, McLean Imaging Center, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-P-001099; Grant # AA10536 (Other Grant/Funding Number: NIAAA)
Record Dates: First submitted 2012-05-09; First posted 2012-05-10 (Estimated); Results first posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Alcohol Consumption
Keywords: Alcohol consumption; Kudzu extract
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): This is a study designed to test whether a single administration of kudzu extract (2 mg) or placebo will significantly reduce the number of drinks consumed during a single 1 ½ hours drinking session when given as a pretreatment 2 ½ hours before the drinking session.
  Interventions: Dietary Supplement: Placebo
- Kudzu (Active Comparator): Kudzu 2mg
  Interventions: Dietary Supplement: Kudzu

INTERVENTIONS:
Dietary Supplement: Kudzu — Kudzu (2 mg) will be administered as a pretreatment 2 ½ hours before a drinking session to see if it will significantly reduce the number of drinks consumed during a single 1 ½ hours drinking session.
  Other Names: Kudzu root extract (NPI-031); Puerariae lobata; Alkontrol-Herbal®
  Arms: Kudzu
Dietary Supplement: Placebo — Placebo will be administered as a pretreatment 2 ½ hours before a drinking session
  Arms: Placebo

SUMMARY:
This is a study designed to test whether a single administration of kudzu extract (2 mg) will significantly reduce the number of drinks consumed during a single 1 ½ hours drinking session when given as pretreatment 2 ½ hours before the drinking session.

DETAILED DESCRIPTION:
In a laboratory experimental setting, subjects will be treated with placebo or 2 grams of kudzu extract 2.5 hours before an afternoon drinking session. The investigators hypothesis is that the kudzu pretreatment will reduce alcohol consumption in this free choice, self-administration paradigm.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding and complying with the protocol
* Good physical and mental health (normal physical exam, ECG, blood and urine chemistries)
* Body Mass Index between 18-30, inclusive
* Age 21-40 years
* Moderate to heavy alcohol drinkers (on the average 20+ drinks/week) or a self-reported pattern of incidences of binge drinking 2 or more times per week (4 or more alcoholic beverages in one sitting)
* Have a stable living situation with current postal address

Exclusion Criteria:

* Concurrent diagnosis of Axis I disorder
* Current or past alcohol dependence; may meet criteria for alcohol abuse. Other drug dependence acceptable only if greater than 3 years.
* Immediate family history pattern of alcoholism or problem drinking (parents or siblings)
* Current drug abuse (other than alcohol or marijuana abuse). Past drug abuse is acceptable.
* Subjects cannot be actively seeking treatment for any drug or alcohol dependence.
* Subjects cannot use marijuana more than once a week. Marijuana abuse/dependence are acceptable if the use criteria is met.
* Maintained on an antipsychotic or antidepressant medication; taking prescription medications except certain short-term anti fungal agents and some tropical creams for dermal conditions.
* Tobacco use greater than 5 cigarettes per day
* History of major head trauma resulting in cognitive impairment or history of seizure disorder
* Heavy caffeine use (greater than 500 mg on a regular, daily basis)
* Subject has active hepatitis and/or aspartate aminotransferase (AST), alanine aminotransferase (ALT) > 3x the upper limit of normal
* For female volunteers, a positive pregnancy test

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-05; Primary Completion 2013-05 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott E. Lukas, Ph.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

REFERENCES:
- [Derived] Penetar DM, Toto LH, Lee DY, Lukas SE. A single dose of kudzu extract reduces alcohol consumption in a binge drinking paradigm. Drug Alcohol Depend. 2015 Aug 1;153:194-200. doi: 10.1016/j.drugalcdep.2015.05.025. Epub 2015 May 27. PMID 26048637
- See also: Related Info — http://www.mclean.harvard.edu/research/neuroimaging/bprl/kudzu.php

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Kudzu
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Kudzu | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.6 (3.3) | 22.6 (3.7) | 23.6 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 10 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 9 | 18
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Drinking Behaviors
Description: A variety of measures describing the drinking behavior will be analyzed with appropriate parametric tests (t-test, analysis of variance): number of beers consumed, weight and volume consumed, sip analysis (number, interlude), and latency (time to open first and subsequent drinks).
Time Frame: Study end
Measure: Mean (Standard Deviation); unit: beers consumed
Groups:
- Placebo: Placebo did not alter alcohol consumption compared to baseline.
- Kudzu: Kudzu extract treatment significantly reduced the number of beers opened and total amounts (weight and volume) consumed. Latency and time to consume a beer was not significantly altered, and there was no difference in the number of sips taken to drink a beer.
Arm/Group | Placebo | Kudzu
Number analyzed (Participants) | 10 | 10
beers consumed | 3.4 (1.1) | 1.9 (1.3)

ADVERSE EVENTS:
Arm/Group | Placebo | Kudzu
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No